CLINICAL TRIAL: NCT03201900
Title: A Multicenter, Uncontrolled, Open-label Study and Extension Study for Verification of Eefficacy and Safety for Perampanel Monotherapy in Untreated Patients With Partial Onset Seizures (Including Secondarily Generalized Seizures) (FREEDOM Study)
Brief Title: Study for Verification of Efficacy and Safety for Perampanel Monotherapy in Untreated Participants With Partial Onset Seizures (Including Secondarily Generalized Seizures (FREEDOM Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-J000-342
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2020-02

CONDITIONS: Partial Onset Seizures
Keywords: perampanel
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- E2007 (Experimental): The Treatment Phase consists of the 4 milligrams (mg) Treatment Phase (the Titration Period [6 weeks] and the Maintenance Period [26 weeks]) and the 8 mg Treatment Phase (the Titration Period [4 weeks] and the Maintenance Period [26 weeks]) if participants require a higher dose. In the 4 mg Titration Period (6 weeks), participants will initiate 2 mg perampanel once daily (QD) for 2 weeks and then will be up-titrated to 4 mg QD and will continue this dose for 4 weeks. If participants have no safety issues at the end of the Titration Period, they will start the 4 mg Maintenance Period for 26 weeks. Participants will only need the higher dose if they are having seizures. In the 8 mg Titration Period (4 weeks), participants will be administered 6 mg perampanel QD for 2 weeks and then will be up-titrated to 8 mg QD and will continue this dose for 2 weeks. If participants have no safety issues at the end of the Titration Period, they will start the 8 mg Maintenance Period for 26 weeks.
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007 — Oral tablet
  Other Names: Perampanel; Fycompa; 2-(2-Oxo-1-phenyl-5-pyridin-2-yl-1,2-dihydropyridin-3-yl) benzonitrile hydrate (4:3)

SUMMARY:
This study is conducted to evaluate the seizure-free rate of the 26-week Maintenance Period in untreated participants with partial onset seizures (POS).

ELIGIBILITY:
Inclusion Criteria:

* Be considered reliable and willing to be available for the study period and are able to record seizures and report adverse events (AEs) himself/herself or have a caregiver who can record seizures and report AEs for them
* Participants who are newly diagnosed or recurrent epilepsy and have experienced at least 2 unprovoked seizures separated by a minimum of 24 hours in the 1 year prior to the Pretreatment Phase
* Participants who have excluded the progressive central nervous system (CNS) abnormality occurring seizures by computed tomography (CT) or magnetic resonance imaging (MRI)
* Participants who have had a diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization-related epilepsy; normal interictal EEGs will be allowed provided that the participant meets the other diagnosis criterion (ie, clinical history)

Exclusion Criteria:

* Participants who present only simple partial seizures without motor signs
* Participants who have seizure clusters where individual seizures cannot be counted
* Participants who present or have a history of Lennox-Gastaut syndrome
* Participants who have a history of status epilepticus
* Participants who have a history of psychogenic non-epileptic seizures
* Participants who have a history of suicidal ideation/attempt
* Participants who present clinically problematic psychological or neurological disorder(s)
* Evidence of clinically significant disease
* Evidence of clinically significant active hepatic disease
* A prolonged time from the beginning of the QRS complex to the end of the T wave (QT) interval corrected for heart rate
* Participants who have a history of receiving any AEDs (except for AEDs used as rescue treatment), antipsychotics or anti-anxiety drugs within 12 weeks prior to the Pretreatment Phase
* Participants who have not used a stable dose of antidepressant in the 12 weeks
* Participants who have a history of any type of surgery for brain or central nervous system within 1 year
* Participants who have a history of receiving any AED (including AED used as rescue treatment) for more than 2 weeks
* Participants who have used intermittent rescue benzodiazepines on 2 or more occasions within 4 weeks
* Participants who have a history of receiving any AED polytherapy
* Participants who experienced treatment with perampanel
* Participants who have had non-constant ketogenic diet within 4 weeks
* Participants who have a history of drug or alcohol dependency or abuse
* Participants who have had multiple drug allergies or a severe drug reaction to an AED(s)
* Females who are breastfeeding or pregnant in the Pretreatment Phase (as documented by a positive beta-human chorionic gonadotropin [β-hCG] test)
* Females of childbearing potential who:

  * Within 28 days before the start of the Pretreatment Phase, did not use a highly effective method of contraception, which includes any of the following:

    * total abstinence (if it is their preferred and usual lifestyle);
    * an intrauterine device or intrauterine hormone-releasing system (IUS);
    * a contraceptive implant;
    * an oral contraceptive (with additional barrier method) (Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation);
    * have a vasectomized partner with confirmed azoospermia
  * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation
* Participants who have participated in a study involving administration of an investigational drug or device within 4 weeks before Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer

Ages: 12 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- Japan (31):
  - Eisai Trial Site #18, Aichi
  - Eisai Trial Site #19, Aichi
  - Eisai Trial Site #11, Fukuoka
  - Eisai Trial Site #29, Fukuoka
  - Eisai Trial Site #4, Hiroshima
  - Eisai Trial Site #16, Hokkaido
  - Eisai Trial Site #8, Hokkaido
  - Eisai Trial Site #14, Hyōgo
  - Eisai Trial Site #6, Hyōgo
  - Eisai Trial Site #7, Kagoshima
  - Eisai Trial Site #9, Kanagawa
  - Eisai Trial Site #10, Kyoto
  - Eisai Trial Site #30, Miyagi
  - Eisai Trial Site #25, Nagasaki
  - Eisai Trial Site #27, Nagasaki
  - Eisai Trial Site #15, Nara
  - Eisai Trial Site #12, Niigata
  - Eisai Trial Site #21, Osaka
  - Eisai Trial Site #24, Osaka
  - Eisai Trial Site #26, Osaka
  - Eisai Trial Site #3, Saitama
  - Eisai Trial Site #5, Saitama
  - Eisai Trial Site #1, Shizuoka
  - Eisai Trial Site #22, Tochigi
  - Eisai Trial Site #28, Tokushima
  - Eisai Trial Site #20, Tokyo
  - Eisai Trial Site #23, Tokyo
  - Eisai Trial Site #31, Tokyo
  - Eisai Trial Site #13, Yamagata
  - Eisai Trial Site #17, Yamaguchi
  - Eisai Trial Site #32, Yamaguchi
- South Korea (7):
  - Eisai Trial Site #38, Gyeonggi-do
  - Eisai Trial Site #36, Incheon
  - Eisai Trial Site # 2, Seoul
  - Eisai Trial Site #33, Seoul
  - Eisai Trial Site #34, Seoul
  - Eisai Trial Site #35, Seoul
  - Eisai Trial Site #37, Seoul

REFERENCES:
- [Derived] Husni RE, Ngo LY, Senokuchi H, Patten A, Hiramatsu H, Watanabe K, Yamamoto T. Experience of perampanel monotherapy beyond initial titration to achieve seizure freedom in patients with focal-onset seizures with newly diagnosed or currently untreated recurrent epilepsy: A post hoc analysis of the open-label Study 342 (FREEDOM). Epilepsia Open. 2022 Mar;7(1):59-66. doi: 10.1002/epi4.12551. Epub 2021 Nov 19. PMID 34657389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 38 investigative sites in Japan and Korea from 28 Jun 2017 to 27 Jul 2020. A total of 98 participants were screened, of which 07 were screen failures and 91 entered Treatment Phase. Of these, 89 participants received the study treatment.
Pre-assignment Details: Study consisted of 2 main phases: Treatment Phase (consisted of a 4 milligram [mg] Treatment Phase [Titration Period {6 weeks} and Maintenance Period {26 weeks}], and for those participants who need a higher dose, the 8 mg Treatment Phase [Titration Period {4 weeks} and Maintenance Period {26 weeks}]) and Extension Phase.
Groups:
- Perampanel: Participants received 2 mg of perampanel tablets orally QD for up to 2 weeks, then dose was up-titrated to 4 mg QD for 4 weeks in 4-mg Titration Period (6 Weeks) followed by 4 mg of perampanel tablets orally QD in Maintenance Period (26 weeks). If a participant experienced seizures during 4-mg Maintenance Period, the participant was transitioned to 8-mg Titration Period based on the participant's safety and tolerability. In 8-mg Titration Period (4 weeks), participants received 6 mg of perampanel tablets orally QD for 2 weeks and up-titrated to 8 mg QD for 2 weeks followed by 8 mg of perampanel tablets orally QD in Maintenance Period (26 weeks). Participants who completed Treatment Phase or who ended Maintenance Period of Treatment Phase due to insufficient efficacy or intolerability, and who agreed to continue perampanel monotherapy entered Extension Phase and received perampanel tablets in 2 mg to 8 mg dose range at the discretion of the investigator based on the participants clinical response and/or tolerability until insufficient seizure control or lack of tolerability, or initiation of additional antiepileptic drug (AEDs).
Period: Treatment Phase (Up to 62 Weeks)
Arm/Group | Perampanel
Started | 91
Treated | 89
Completed | 54
Not Completed | 37
Not completed — Adverse Event | 9
Not completed — Subject Choice | 1
Not completed — Inadequate therapeutic effect | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal of consent | 6
Not completed — Other than specified | 11
Not completed — Not treated | 2
Period: Extension Phase (From Week 63 to 156)
Arm/Group | Perampanel
Started | 46 (Eligible participants who completed Treatment Phase and agreed to continue in the Extension Phase.)
Completed | 38
Not Completed | 8
Not completed — Subject choice | 1
Not completed — Pregnancy | 1
Not completed — Inadequate therapeutic effect | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal of consent | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who signed informed consent, received at least 1 dose of study drug and had at least one post dose safety assessment.
Groups:
- Perampanel: Participants received 2 mg of perampanel tablets orally QD for up to 2 weeks, then dose was up-titrated to 4 mg QD for 4 weeks in 4-mg Titration Period (6 Weeks) followed by 4 mg of perampanel tablets orally QD in Maintenance Period (26 weeks). If a participant experienced seizures during 4-mg Maintenance Period, the participant was transitioned to 8-mg Titration Period based on the participant's safety and tolerability. In 8-mg Titration Period (4 weeks), participants received 6 mg of perampanel tablets orally QD for 2 weeks and up-titrated to 8 mg QD for 2 weeks followed by 8 mg of perampanel tablets orally QD in Maintenance Period (26 weeks). Participants who completed Treatment Phase or who ended Maintenance Period of Treatment Phase due to insufficient efficacy or intolerability, and who agreed to continue perampanel monotherapy entered Extension Phase and received perampanel tablets in 2 mg to 8 mg dose range at the discretion of the investigator based on the participants clinical response and/or tolerability until insufficient seizure control or lack of tolerability, or initiation of AEDs.
Arm/Group | Perampanel
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (18.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 89
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Partial-onset Seizures (POS) Who Achieved Seizure-free Status During the 26-week Maintenance Period of 4 mg Perampanel
Description: A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. POS was a seizure that starts in one area of the brain that may or may not associated with loss of awareness and consciousness. Seizure-free status was defined as no incidence of seizure during 26-week Maintenance Period of 4 mg perampanel.
Time Frame: 26 weeks in Maintenance Period of 4 mg perampanel
Population: Modified intent to treat (mITT) set: group of participants who signed informed consent, received at least 1 dose of study drug, who entered the 4-mg Maintenance Period and had at least 1 postdose primary efficacy measurement in the 26-week Maintenance Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 73
percentage of participants | 63.0 [50.9 to 74.0]

2. Secondary Outcome: Percentage of Participants With POS Who Achieved Seizure-free Status During the 26-week Maintenance Period of Last Evaluated Dose of 4 or 8 mg Perampanel
Description: A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. POS was a seizure that starts in one area of the brain that may or may not associated with loss of awareness and consciousness. Seizure-free status was defined as no incidence of seizure during the 26-week Maintenance Period of last evaluated dose of 4 or 8 mg perampanel.
Time Frame: 26 weeks in Maintenance Period of 4 or 8 mg perampanel
Population: mITT set: group of participants who signed informed consent, received at least 1 dose of study drug, who entered the 4-mg Maintenance Period and had at least 1 postdose primary efficacy measurement in the 26-week Maintenance Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 73
percentage of participants | 74.0 [62.4 to 83.5]

3. Secondary Outcome: Percentage of Participants With POS Who Achieved Seizure-free Status During the 52-week Treatment Phase (26-week Maintenance Period Plus 26-week Extension Phase) of 4 mg of Perampanel
Description: A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. POS was a seizure that starts in one area of the brain that may or may not associated with loss of awareness and consciousness. Seizure-free status was defined as no incidence of seizure during 52-weeks treatment of 4 mg perampanel.
Time Frame: 52-week (Maintenance Period of 4 mg perampanel + Extension Phase of 4 mg perampanel)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 73
percentage of participants | 32.9 [22.3 to 44.9]

4. Secondary Outcome: Percentage of Participants With POS Who Achieved Seizure-free Status During the 52-week of Treatment Phase (26-week Maintenance Period Plus 26-week Extension Phase) of Last Evaluated Dose of 4 or 8 mg Perampanel
Description: A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. POS was a seizure that starts in one area of the brain that may or may not associated with loss of awareness and consciousness. Seizure-free status was defined as no incidence of seizure during the 52-week treatment of last evaluated dose of 4 or 8 mg perampanel.
Time Frame: 52-week (Maintenance Period of last evaluated dose of 4 or 8 mg perampanel + Extension Phase of 4 or 8 mg perampanel)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 73
percentage of participants | 42.5 [31.0 to 54.6]

5. Secondary Outcome: Time to Onset of First Seizure From the First Dose of Study Drug in the Maintenance Period of 4 mg Perampanel
Description: Time to onset of first seizure was defined as the period from the first dose of study drug in the 4 mg Maintenance Period to the onset of first seizure. A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain.
Time Frame: From the first dose of study drug in the Maintenance Period (Week 6) up to the first seizure onset (up to 150 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Perampanel
Number analyzed (Participants) | 73
weeks | NA [37.4 to NA] — Median and upper 95% CI value was not estimable because less than (<) 50 percent (%) of participants experienced a POS seizure event.

6. Secondary Outcome: Time to Onset of First Seizure From the First Dose of Study Drug in the Maintenance Period of Last Evaluated Dose of 4 or 8 mg Perampanel
Description: Time to onset of first seizure was defined as the period from the first dose of study drug in the 4 mg or 8 mg Maintenance Period to the onset of first seizure. A seizure was a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain.
Time Frame: From the first dose of study drug in the Maintenance Period (Week 6) up to the first seizure onset (up to 150 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Perampanel
Number analyzed (Participants) | 73
weeks | NA [NA to NA] — Median, upper and lower 95% CI value was not estimable because <50% of participants experienced a POS seizure event.

7. Secondary Outcome: Time to Withdrawal From the First Dose of Study Drug in the Maintenance Period of 4 mg Perampanel
Description: Time to withdrawal from the study was defined as the period from the first dose of study drug in the 4 mg Maintenance Period to the date of withdrawal from study, regardless of reason.
Time Frame: From the first dose of study drug in the Maintenance Period (Week 6) up to the date of first withdrawal, regardless of reason (up to 150 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Perampanel
Number analyzed (Participants) | 73
weeks | NA [27.4 to NA] — Median and upper 95% CI value was not estimable because <50% of participants discontinued the study.

8. Secondary Outcome: Time to Withdrawal From the First Dose of Study Drug in the Maintenance Period of Last Evaluated Dose of 4 or 8 mg Perampanel
Description: Time to withdrawal from the study was defined as the period from the first dose of study drug in the 4 mg or 8 mg Maintenance Period to the date of withdrawal from study, regardless of reason.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Perampanel
Number analyzed (Participants) | 73
weeks | NA [27.4 to NA] — Median and upper 95% CI value was not estimable because <50% of participants discontinued the study.

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Event (TESAEs), and TEAEs Leading to Discontinuation of the Study Drug
Time Frame: From baseline up to 28 days after last dose of study drug (up to 160 weeks)
Population: The safety analysis set was the group of participants who signed informed consent, received at least one dose of study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Perampanel
Number analyzed (Participants) | 89
Participants
  TEAEs | 74
  TESAEs | 13
  TEAEs leading to discontinuation of study drug | 9

ADVERSE EVENTS:
Time Frame: From baseline up to 28 days after last dose of study drug (up to 160 weeks)
Arm/Group | Perampanel
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 13/89
Other Adverse Events (participants affected / at risk) | 73/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel (N=89)
Malaise (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (4)
Headache (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel (N=89)
Auditory disorder (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Toothache (Gastrointestinal disorders) | 3 (7)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Feeling abnormal (General disorders) | 4 (4)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 19 (42)
Influenza (Infections and infestations) | 2 (2)
Angular cheilitis (Infections and infestations) | 1 (1)
Enterocolitis viral (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media chronic (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1)
Trichophytosis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 4 (4)
Weight increased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 34 (40)
Somnolence (Nervous system disorders) | 12 (13)
Headache (Nervous system disorders) | 12 (15)
Epilepsy (Nervous system disorders) | 4 (4)
Amnesia (Nervous system disorders) | 2 (2)
Hypersomnia (Nervous system disorders) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Postictal headache (Nervous system disorders) | 1 (4)
Syncope (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Irritability (Psychiatric disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Affect lability (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Emotional disorder (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Posterior capsule opacification (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gingival atrophy (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT03201900/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03201900/SAP_001.pdf